CLINICAL TRIAL: NCT06323707
Title: Implementing Physical Activity for Individuals With Cancer During Treatment: The IMPACT Implementation-Effectiveness Trial
Brief Title: The IMPACT Implementation-Effectiveness Trial
Acronym: IMPACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Hamilton Health Sciences Corporation (Other); Niagara Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IMPACT
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise & Self-Management (Experimental)
  Interventions: Behavioral: Exercise; Behavioral: Self-management e-module
- Self-Management Only (Experimental)
  Interventions: Behavioral: Self-management e-module
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — Eight sessions of moderate intensity aerobic exercise using recumbent bike within the cancer institution.
  Arms: Exercise & Self-Management
Behavioral: Self-management e-module — Eight 15 minute self-management e-modules related to exercise and physical activity for cancer survivors.
  Arms: Exercise & Self-Management; Self-Management Only

SUMMARY:
More Canadians are surviving cancer, however, individuals with cancer live with side effects for years after treatments have ended. The physical and psychosocial benefits of regular physical activity (PA) during and after cancer treatment are well established. However, less than 30% of individuals with cancer meet current PA recommendations and PA levels decline significantly during treatment. PA services within the cancer institution to support well-being during treatment are not available for survivors across Ontario. Strategies are needed within cancer centres to close the gap between the evidence and clinical practice.

What is the purpose? To evaluate the effectiveness of a novel exercise and education strategy for individuals with cancer during treatment.

What are we proposing to do? This project includes two parts. In Part 1 participants will be put into one of three groups. Group 1 (Exercise & self-management) will include eight sessions of supervised, institution-based exercise and self-management education. Group 2 (self-management only) will include eight virtual self-management education sessions with an exercise professional. Group 3 will receive usual care (i.e., no intervention).

In Part 2 participants who attended less than 75% of their sessions will be asked to complete an interview on the barriers to continuing with the study during cancer treatment.

Why is this work important? Findings from this trial will inform the way PA services are provided within cancer institutions across Ontario. This novel strategy incorporates both institution-based and home-based exercise strategies during treatment and highlights the importance of individuals with cancer taking an active role in managing their condition during treatment. This can prevent future complications and decrease burden on the individual and the healthcare system. Results will inform future decisions on PA implementation strategies for cancer survivors with diverse needs across Ontario.

DETAILED DESCRIPTION:
Rationale:

The burden of cancer in Canada is growing. More individuals are surviving cancer, however, individuals with cancer live with side effects for years after treatments have ended. The physical and psychosocial benefits of regular physical activity (PA) during and after cancer treatment are well established. However, less than 30% of individuals with cancer meet current PA recommendations and PA levels decline significantly during active treatment. Institution-based PA services to support wellbeing and minimize burden during treatment are not available across Ontario. Novel implementation strategies are needed within the institution to close the gap between the evidence and clinical practice. Implementation research allows us to understand how to deliver interventions effectively in diverse settings.

Aim & Objectives:

The overall aim of this project is to conduct a fully powered, multi-centred randomized controlled trial (RCT) to evaluate the effectiveness of a novel implementation strategy including exercise and SM versus usual care for individuals with cancer during treatment. To do this, there are two main objectives: 1) Determine the feasibility and effectiveness of a novel implementation strategy using exercise and SM during treatment

Methods:

Study Design: Effectiveness-Implementation RCT Participants: Adults (>18 years) with a cancer diagnosis of any stage, currently receiving treatment, and cleared for exercise by their oncology care team will be included in this study.

Procedure: Participants will be randomized to three groups. Group 1: Exercise & SM: Eight sessions of supervised, in-person institution-based exercise and SM education. This group will also receive 4 booster sessions by telephone post intervention.

Group 2: SM Only: Eight virtual sessions of SM education using video conferencing with a qualified exercise professional. This group will also receive 4 booster sessions by phone post intervention.

Group 3: Usual care: No intervention.

Significance:

Implementation research is crucial to improving our understanding of real-world factors that impact successful application of research in healthcare settings. This novel implementation strategy builds off previous work and incorporates institution-based exercise and SM during treatment. Findings from this trial will build off our previous work and inform the way PA services are provided within cancer institutions across Ontario. Our goal is to make these services available to all individuals with cancer during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. adults with a cancer diagnosis (any type or stage)
2. individuals are currently receiving treatment for cancer
3. individuals have been cleared for exercise by their oncology care team

Exclusion Criteria:

1) Self-report any chronic condition, cognitive impairment, or injury that would prevent them from participating in moderate intensity exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | 16-weeks
  Godin Leisure Time Exercise Questionnaire
Physical activity level | 12-months
  Godin Leisure Time Exercise Questionnaire
Physical activity level | 6-months
  Godin Leisure Time Exercise Questionnaire

SECONDARY OUTCOMES:
Quality of life | 16-weeks
  Measured using the Functional Assessment of Cancer Therapy-General (FACT-G). Total scores range from 0-108 with higher scores representing higher quality of life.
Quality of life | 6-months
  Measured using the Functional Assessment of Cancer Therapy-General (FACT-G). Total scores range from 0-108 with higher scores representing higher quality of life.
Quality of life | 12-months
  Measured using the Functional Assessment of Cancer Therapy-General (FACT-G). Total scores range from 0-108 with higher scores representing higher quality of life.
Level of exercise knowledge | 16-weeks
  Measured using the 'Theory of Planned Behaviour Questionnaire'. Total scores range from 8-56 with higher scores representing higher levels of exercise knowledge.
Level of exercise knowledge | 6-months
  Measured using the 'Theory of Planned Behaviour Questionnaire'. Total scores range from 8-56 with higher scores representing higher levels of exercise knowledge.
Level of exercise knowledge | 12-months
  Measured using the 'Theory of Planned Behaviour Questionnaire'. Total scores range from 8-56 with higher scores representing higher levels of exercise knowledge.
Health status | 16-weeks
  Measured using the Eq-5d-3L VAS. Measured on a scale of 0-100 with higher scores representing higher levels perceived health status.
Health status | 6-months
  Measured using the Eq-5d-3L VAS. Measured on a scale of 0-100 with higher scores representing higher levels perceived health status.
Health status | 12-months
  Measured using the Eq-5d-3L VAS. Measured on a scale of 0-100 with higher scores representing higher levels perceived health status.
Aerobic capacity | 16-weeks
  Six minute walk test
Aerobic capacity | 6-months
  Six minute walk test
Aerobic capacity | 12-months
  Six minute walk test
Cardiovascular outcomes - Blood pressure | 16-weeks
  Resting Blood Pressure
Cardiovascular outcomes - Blood pressure | 6-months
  Resting Blood Pressure
Cardiovascular outcomes - Blood pressure | 12-months
  Resting Blood Pressure
Cardiovascular outcomes - Heart rate | 16-weeks
  Resting heart rate
Cardiovascular outcomes - Heart rate | 6-months
  Resting heart rate
Cardiovascular outcomes - Heart rate | 12-months
  Resting heart rate

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Joseph Brant Hospital, Burlington, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Walker Family Cancer Centre, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith-Turchyn J, Sabiston CM, Edward H, Richardson J, Nayiga BK, Page A, Brooks D, Mukherjee SD. Implementing physical activity for individuals with cancer during treatment: protocol for the IMPACT implementation-effectiveness trial. BMJ Open. 2025 Mar 27;15(3):e101013. doi: 10.1136/bmjopen-2025-101013. PMID 40148001